CLINICAL TRIAL: NCT02237092
Title: Effect of Intra-abdominal Pressure to the Level of the Sensory Block at Caesarean Section Under Spinal Anesthesia
Acronym: IAPSB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tver Regional Perinatal Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TR-1
Record Dates: First submitted 2014-09-02; First posted 2014-09-11 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Obstetric Anesthesia Problems; High-Risk Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Measurement of IAP (Experimental): The data obtained are in inches of water column were translated in millimeters of mercury.
  Interventions: Procedure: Measurement of IAP

INTERVENTIONS:
Procedure: Measurement of IAP — The level of intra-abdominal pressure was measured via a Foley catheter through the urinary bladder. After the introduction of a 30 mL of warm saline. Measurement of the water column in the system was made from the zero level to the mid-axillary line, for 10 minutes, after quiet breathing pregnant at the time of expiration.

SUMMARY:
It is known that an increase in intra-abdominal pressure (IAP) causes a decrease in the volume of cerebrospinal fluid in the lumbar and lower thoracic region, which may contribute to the development of more high spinal block.

DETAILED DESCRIPTION:
There is a hypothesis, the higher the level of intra-abdominal pressure, the greater the likelihood of developing a high-level (=>Th4) sensor block.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 36 - 40 weeks
* Singleton pregnancies
* Elective caesarean section

Exclusion Criteria:

* Gestational age <= 35 weeks
* Twins pregnancies
* Disease the cardiovascular system (hypertension, etc.)
* Non-elective caesarean section

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandr Ronenson, PhD student, Principal Investigator — Tver Regional Perinatal Center; Sergei Sitkin, DMedSc, Study Director — Tver State Medical Academy
Locations (1):
- Tver Regional Perinatal Center, Tver', Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] S. Sitkin, A. Ronenson, J. Savelieva, M. Cherdyntsev. Prediction of high level spinal block in caesarean section. Regional Anesthesia and Pain Medicine. - 2012. - Volume 37. - Sup 1 5. - p. 183.
- [Result] Sitkin, S.; Ronenson, A.; Wagle, S.; Saveleva, J. Effect of intra-abdominal pressure of pregnancy for the development of spinal block for cesarean section: 11AP1-10. European Journal of Anaesthesiology. - 2013 - Volume 30. - Sup 51. - p. 167-168.
- [Result] Sitkin S., Ronenson A.M., Savelieva J.V., Wagle S. Influence of intra-abdominal pressure (iap) and body mass index (bmi) in pregnancy on the development of spinal block for cesarean section. Regional Anesthesia and Pain Medicine, Volume 38, Number 5, Supplement 1 5, September-October. - 2013. - p. 179
- See also: Patent on the research — http://www.freepatent.ru/images/patents/497/2499554/patent-2499554.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Gestational age 36 - 40 weeks, Singleton pregnancies, Elective caesarean section
Period: Overall Study
Arm/Group | Measurement of IAP
Started | 196
Completed | 196
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Pregnant planned for cesarean section
Groups:
- Measurement of IAP: Measurement of IAP: The level of intra-abdominal pressure was measured via a Foley catheter through the urinary bladder. After the introduction of a 30 mL of warm saline. Measurement of the water column in the system was made from the zero level to the mid-axillary line, for 10 minutes, after quiet breathing pregnant at the time of expiration.The data obtained are in inches of water column were translated in millimeters of mercury.
Arm/Group | Measurement of IAP
Number analyzed (Participants) | 196
Age, Continuous [Median (Standard Deviation); unit: years] | 29.5 (5.7)
Sex/Gender, Customized [Number; unit: Pregnant women]
  Female | 196
  Male | 0
Height [Median (Standard Deviation); unit: cm] | 163.9 (7.4)
Body mass index [Median (Standard Deviation); unit: kg/m^2] | 30.8 (5.7)
Abdominal circumference [Median (Standard Deviation); unit: cm] | 105.1 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: The Level of Intra-abdominal Pressure (IAP)
Description: Measurement of IAP: The level of intra-abdominal pressure was measured via a Foley catheter through the urinary bladder. After the introduction of a 30 mL of warm saline. Measurement of the water column in the system was made from the zero level to the mid-axillary line, after quiet breathing pregnant at the time of expiration. The data obtained are in inches of water column were translated in millimeters of mercury.
Time Frame: Before spinal anesthesia, average 10 minutes.
Measure: Median (Standard Error); unit: mm Hg
Groups:
- Intra-abdominal Pressure (IAP) in Pregnant Women: Average IAP in pregnant women
Arm/Group | Intra-abdominal Pressure (IAP) in Pregnant Women
Number analyzed (Participants) | 196
mm Hg | 15.33 (0.17)

2. Primary Outcome: Classification Grade of Intra-abdominal Hypertension (IAH)
Description: Average IAP in pregnant women with different Grade of intra-abdominal hypertension Physiological norm (≤11,99 mm Hg) Grade I (12 - 15.99 mm Hg) Grade II (16 - 20.99 mm Hg) Grade III (21 - 25.99 mm Hg)
Time Frame: Before spinal anesthesia, average 10 minutes.
Measure: Median (Standard Error); unit: mm Hg
Groups:
- Physiological Norm: (≤11,99 mm Hg)
- Grade I: (12 - 15.99 mm Hg)
- Grade II: (16 - 20.99 mm Hg)
- Grade III: (21 - 25.99 mm Hg)
Arm/Group | Physiological Norm | Grade I | Grade II | Grade III
Number analyzed (Participants) | 18 | 96 | 79 | 3
mm Hg | 11.60 (0.09) | 14.11 (0.10) | 17.43 (0.14) | 21.56 (0.25)

3. Secondary Outcome: Level of Sensory Blocks
Description: Block level of thoracic vertebrae are reported for pregnant women who had level of sensory block higher than 4 thoracic vertebra and less than 5 thoracic vertebra
Time Frame: After spinal anesthesia, average 20 minutes.
Measure: Median (Standard Error); unit: Block level level of thoracic vertebrae
Groups:
- Level of Sensory Block => Th4 (Spinal Anesthesia); Level of Sensory Block < = Th5 (Spinal Anesthesia): Pregnant with the level of sensory block in 20 minutes after the start of spinal anesthesia
Arm/Group | Level of Sensory Block => Th4 (Spinal Anesthesia) | Level of Sensory Block < = Th5 (Spinal Anesthesia)
Number analyzed (Participants) | 62 | 134
Block level level of thoracic vertebrae | 3.5 (0.1) | 5.8 (0.1)
Statistical Analysis 1: Comparison: Level of Sensory Block => Th4 (Spinal Anesthesia) vs Level of Sensory Block < = Th5 (Spinal Anesthesia); Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Obesity and IAP
Description: Effect of obesity on the level of IAP
Time Frame: Before spinal anesthesia, average 10 minutes.
Measure: Median (Standard Error); unit: mm Hg
Groups:
- No Obesity: BMI < = 29.99
- Obesity: BMI = > 30.00
Arm/Group | No Obesity | Obesity
Number analyzed (Participants) | 98 | 98
mm Hg | 14.61 (0.20) | 16.06 (0.25)
Statistical Analysis 1: Comparison: No Obesity vs Obesity; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: The Level of IAP
Description: The level of IAP in obstetric patients in the groups with high ( => Th4) and low (< = Th5) blocks
Time Frame: After spinal anesthesia, average 20 minutes.
Measure: Median (Standard Error); unit: mm Hg
Arm/Group | Level of Sensory Block => Th4 (Spinal Anesthesia) | Level of Sensory Block < = Th5 (Spinal Anesthesia)
Number analyzed (Participants) | 62 | 134
mm Hg | 16.5 (0.3) | 14.0 (0.2)
Statistical Analysis 1: Comparison: Level of Sensory Block => Th4 (Spinal Anesthesia) vs Level of Sensory Block < = Th5 (Spinal Anesthesia); Test type: Superiority or Other; p < 0.02, t-test, 2 sided

6. Secondary Outcome: Number of Pregnants With Blocks = > Th4 With IAP Higher or Less Than 16 mm Hg
Time Frame: After spinal anesthesia, average 20 minutes.
Measure: Number; unit: Number of pregnants with Blocks = > Th4
Groups:
- Level of IAP < 16 mm Hg: number of pregnant women with Level of IAP < 16 mm Hg
- Level of IAP = > 16 mm Hg: number of pregnant women with Level of IAP = > 16 mm Hg
Arm/Group | Level of IAP < 16 mm Hg | Level of IAP = > 16 mm Hg
Number analyzed (Participants) | 114 | 82
Number of pregnants with Blocks = > Th4 | 29 | 33
Statistical Analysis 1: Comparison: Level of IAP < 16 mm Hg vs Level of IAP = > 16 mm Hg; Test type: Superiority or Other; p < 0.05, NNT; Risk Ratio (RR) = 1.58, 95% CI 2-sided [1.05 to 2.58]

ADVERSE EVENTS:
Time Frame: During the operation, an average of 30 minutes
Description: Decrease in systolic blood pressure below 90 mm Hg or more than 30% of the base line level of systolic blood pressure
Groups:
- Level of Sensory Block => Th4 (Spinal Anesthesia); Level of Sensory Block < = Th5 (Spinal Anesthesia): Hypotension: Decrease in systolic blood pressure below 90 mm Hg or more than 30% of the base line level of systolic blood pressure
Arm/Group | Level of Sensory Block => Th4 (Spinal Anesthesia) | Level of Sensory Block < = Th5 (Spinal Anesthesia)
Serious Adverse Events (participants affected / at risk) | 23/62 | 17/134
Other Adverse Events (participants affected / at risk) | 0/62 | 0/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level of Sensory Block => Th4 (Spinal Anesthesia) (N=62) | Level of Sensory Block < = Th5 (Spinal Anesthesia) (N=134)
Hypotension (Cardiac disorders) | 23 (23) | 17 (17) — Decrease in systolic blood pressure below 90 mm Hg or more than 30% of the base line level of systolic blood pressure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level of Sensory Block => Th4 (Spinal Anesthesia) (N=62) | Level of Sensory Block < = Th5 (Spinal Anesthesia) (N=134)
Changing the type of anesthesia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) — Changing the type of anesthesia to General anesthesia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes